CLINICAL TRIAL: NCT04941976
Title: Phase IV Study Comparing the Efficacy and Safety of Benzydamine Hydrochloride 0,3% Oromucosal Spray and Benzydamine Hydrochloride 3 mg Lozenges in Patients With Acute Sore Throat
Brief Title: Benzydamine in Sore Throat Pain Relief (BePaiR Study)
Acronym: BePaiR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Zak-Pharma Dienstleistung Ges.m.b.H. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030(Z)WO19176; 2019-003257-29 (EudraCT Number)
Record Dates: First submitted 2021-06-23; First posted 2021-06-28 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Acute Sore Throat
Keywords: oromucosal spray; lozenges; Benzydamine hydrochloride 0.3%; Benzidamine hydrochloride 3 mg; acute sore throat
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Intervention Model Description: Multicenter, randomised, active-controlled, open label, parallel-group, international study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.3% benzydamine hydrochloride spray oromucosal solution (Experimental): A single application of 0.3% benzydamine hydrochloride spray oromucosal solution, corresponding to 2.04 mg of benzydamine (4 nebulizations)
  Interventions: Drug: 0.3% benzydamine hydrochloride spray oromucosal solution
- 3 mg lozenge of benzydamine hydrochloride (mint flavour), corresponding to 2.68 mg of benzydamine (Active Comparator): A single 3 mg lozenge of benzydamine hydrochloride (mint flavour), corresponding to 2.68 mg of benzydamine.
  Interventions: Drug: Single 3 mg lozenge of benzydamine hydrochloride (mint flavour)

INTERVENTIONS:
Drug: 0.3% benzydamine hydrochloride spray oromucosal solution — Single application of 0.3% benzydamine hydrochloride spray oromucosal solution. Drug applications will be performed at the investigational site, on the morning of Visit 0.
  In case of persistent sore throat patients will continue the assigned treatment at home, according to the local SmPC and up to one week, until the symptoms' resolution.
  Arms: 0.3% benzydamine hydrochloride spray oromucosal solution
Drug: Single 3 mg lozenge of benzydamine hydrochloride (mint flavour) — Single 3 mg lozenge of benzydamine hydrochloride (mint flavour). Drug applications will be performed at the investigational site, on the morning of Visit 0.
  In case of persistent sore throat patients will continue the assigned treatment at home, according to the local SmPC and up to one week, until the symptoms' resolution.
  Arms: 3 mg lozenge of benzydamine hydrochloride (mint flavour), corresponding to 2.68 mg of benzydamine

SUMMARY:
The aim of this study is to generate new clinical data about the speed of relief provided by a single application of Benzydamine hydrochloride 0,3% oromucosal spray vs Benzydamine hydrochloride 3 mg lozenges mint flavour.

DETAILED DESCRIPTION:
The efficacy and safety of benzydamine local-applied, in the treatment of various throat inflammatory and painful conditions, had been widely demonstrated.

The aim of this study is to generate new clinical data about the speed of relief provided by a single application of Benzydamine hydrochloride 0,3% oromucosal spray or Benzydamine hydrochloride 3 mg lozenges mint flavour.

The study will be conducted at 15 sites located among Poland, Hungary and Russia (5 sites for each country).

356 patients affected by acute sore throat will be enrolled in out-patient clinics or out-patient departments of city hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients (aged 18 - 75 years, limits included) with recent onset (≤3 days) of sore throat and a diagnosis of tonsillopharyngitis confirmed by:

  1. Presence of at least one symptom of URTI in the previous 24 h on the URTI questionnaire;
  2. Sore throat pain intensity score ≥ 60 mm on Sore Throat Pain Intensity Scale (STPIS);
  3. A score ≥ 5 on Tonsillo-Pharingytis Assessment (TPA);
* Women of childbearing potential or with no menses for a period < 12 months must have a negative pregnancy test at Visit 0 and have to agree not to start a pregnancy from the signature of the informed consent up to the Visit 2, using an appropriate birth control method such as combined oestrogen-progestin containing hormonal contraceptives (e.g., oral, injectable, transdermal), progestin-only hormonal contraceptives (e.g., oral, injectable, implantable), intrauterine device (IUD) or Intrauterine hormone-releasing System (IUS) in combination with male condom, bilateral tubal occlusion, vasectomised partner, sexual abstinence. The following definitions will be considered:

  * Woman of childbearing potential (WOCBP): i.e., fertile, following menarche and until becoming post-menopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
* Patients legally capable of giving their consent to participate in the study (including personal data processing) and available to sign and date the written informed consent.

Exclusion Criteria:

* Known hypersensitivity to benzydamine or its excipients;
* Phenylketonuria;
* Clinically significant abnormalities at physical examination and vital signs;
* Intolerance to acetylsalicylic acid or other NSAIDS;
* History or diagnosis of asthma;
* Any concomitant disease that compromise breathing (i.e. bronchopneumonia);
* Mouth breathing due to nasal congestion which causes throat drying;
* Severe coughing which causes throat discomfort;
* Purulent plaques on the tonsils;
* Any inhaled therapy in the previous week before the first drug administration;
* Use of antibiotics for an acute disease in the 7 days before randomisation (chronic antibiotic use, such as for acne, is acceptable); any sustained release analgesic within 24 hours of administration of study medication; any medications for cold and flu (i.e., decongestants, antihistamines, expectorants, antitussives), immediate release analgesic or antipyretic within 4 hours of administration of study medication;
* Use of any lozenge, mouthwash, spray or menthol-containing products within 2 hours of administration of study medication;
* Women during pregnancy or lactation period;
* Subject involved in the conduct of the study (e.g. Investigator or his/her deputy, first grade relatives, pharmacist, assistant or other personnel, etc);
* Participation to a clinical trial within 3 months prior to the inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of responders at 2 min | 2 minutes
  Percentage of responders defined as patients reported at least a "slight relief" using Sore Throat Relief Rating Scale at 2 minutes after the first application of benzydamine hydrochloride 0.3% spray or benzydamine hydrochloride 3mg lozenges.
  A score ≥1 in Sore Throat Relief Rating Scal is considered as the first perceived pain relief or "slight relief".

SECONDARY OUTCOMES:
Percentage of responders at 1 min | 1 minute
  Percentage of responders defined as patients reported at least a "slight relief" using Sore Throat Relief Rating Scale at 1 minute after the first application of benzydamine hydrochloride 0.3% spray or benzydamine hydrochloride 3mg lozenges.
  A score ≥1 in Sore Throat Relief Rating Scal is considered as the first perceived pain relief or "slight relief".
Percentage of patients recording a meaningful sore throat relief | 5,10,15,30,60 and 120 minutes
  The meaningful sore throat relief is assessed after a single dose administration.
  A "meaningful sore throat relief" is considered as a score ≥ 3 (moderate relief) in the Sore Throat Relief Rating Scale.
Change in Sore Throat Relief Rating Scale. | 1, 2, 5,10,15,30,60,120,240 minutes
  Change from 1 minute up to 4 hours post-dose in Sore Throat Relief Rating Scale.The Sore Throat Relief Rating Scale is a 7-point categorical scale that assesses the local analgesic effect starting from: 0= "no relief" up t 7="complete relief"
Change in sore throat pain intensity. | Baseline, 7 day
  Change in sore throat pain intensity from baseline up to 7 days of treatment through the Sore Throat Pain Intensity Scale assessment. The Sore Throat Pain Intensity Scale is a visual analogic scale (VAS) assessing the intensity of the Sore Throat. It consists of a continuous horizontal line of 100 mm in length with ends labelled as the extremes of pain, from 0 (left side): "no pain", to 10 (right side): "pain as bad as it could be".

CONTACTS AND LOCATIONS:
Locations (15):
- Hungary (4):
  - Háziorvosi Rendelő, Budapest
  - Háziorvosi Rendelő, Érd
  - Háziorvosi Rendelő, Pilisvörösvár
  - Háziorvosi Rendelő, Tárnok
- Poland (5):
  - NZOZ Centrum Zdrowia i Profilaktyki Dabie Filia, Krakow
  - NZOZ Centrum Zdrowia i Profilaktyki Dabie Krakow, Krakow
  - ValeoMedical, Lodz
  - Zdrowa Rodzina Przychodnia Lekarska, Warsaw
  - Przchodnia Orlik, Warsaw
- Russia (6):
  - Scientific research center Eco-Safety, LLC, Saint Petersburg
  - Private Healthcare Institution "Clinical Hospital "RZD-Medicine" St.Petersburg", Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "City outpatient clinic #106", Saint Petersburg
  - Hospital "OrKli" LLC, Saint Petersburg
  - "Astarta" LLC, Saint Petersburg
  - "Meili" LLC, Saint Petersburg